CLINICAL TRIAL: NCT02321579
Title: The Effects of Vitamin B-6 and Glutathione on Inflammatory Responses, Homocysteine Metabolism, Oxidative Stress and Antioxidant Capacities in Patients With Liver Cirrhosis or Hepatocellular Carcinoma
Brief Title: Vitamin B-6 and Glutathione on Inflammation, Homocysteine, Oxidative Stress and Antioxidant Capacities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SF14261B
Record Dates: First submitted 2014-12-09; First posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Liver Cirrhosis; Liver Cancer
MeSH Terms: conditions — Liver Cirrhosis; Liver Neoplasms | interventions — Vitamin B 6; Glutathione; Dextrins

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Negative control (Placebo Comparator): Dextrins
  Interventions: Dietary Supplement: Dextrins
- Supplement 1 (Experimental): 50 mg/d vitamin B-6
  Interventions: Dietary Supplement: vitamin B-6
- Supplement 2 (Experimental): 500 mg/d Glutathione
  Interventions: Dietary Supplement: Glutathione
- Supplement 3 (Experimental): 50 mg/d vitamin B-6 plus 500 mg/d Glutathione
  Interventions: Dietary Supplement: vitamin B-6; Dietary Supplement: Glutathione

INTERVENTIONS:
Dietary Supplement: vitamin B-6 — 50 mg/d
  Arms: Supplement 1; Supplement 3
Dietary Supplement: Glutathione — 500 mg/d
  Arms: Supplement 2; Supplement 3
Dietary Supplement: Dextrins — 50 mg/d
  Arms: Negative control

SUMMARY:
This study is designed as a hospital-based cross-sectional and randomized placebo-controlled intervention trial. One hundred and fifty patients with either cirrhosis or cirrhosis combined with hepatocellular carcinoma (HCC) who meet the inclusion criteria will be recruited from Taichung General Veterans Hospital. One hundred patients will be randomly assigned to either the 1) placebo group (n = 25); 2) vitamin B-6 group; (50 mg/d, n = 25); 3) glutathione (GSH) group (500 mg/d, n = 25); or 4) vitamin B-6 (50 mg/d) plus GSH (500 mg/d) group (n = 25) for 3 mo. Data on demography, anthropometry and medical history will be collected. Patients with cirrhosis or cirrhosis combined with HCC will have fasting blood drawn in the clinics. Additionally, patients who participated in the intervention study will have blood drawn at month 0, 1, 2 and 3 during intervention period. Hematological measurements, plasma vitamin B-6 status, GSH, inflammatory markers, homocysteine, cysteine, SAM, SAH, oxidative stress indicator, oxidized GSH and GSH related antioxidant enzyme activities will be analyzed.

DETAILED DESCRIPTION:
Liver cirrhosis is now the ninth leading cause of death and hepatocellular carcinoma (HCC) is the second leading cause of cancer mortality among men and women in Taiwan. Vitamin B-6 and glutathione (GSH) are metabolized in liver, the role of vitamin B-6 and GSH playing in the inflammatory responses and antioxidant function would be impaired during hepatic injury. The purpose of this study is going to assess the effects of individual or combined supplementation of vitamin B-6 and GSH on homocysteine, cysteine, the ratio of S-adenosylmethionine (SAM)/S-adenosylhomocysteine (SAH), oxidative stress, oxidized glutathione (GSSG) and GSH related antioxidant enzyme activities in patients with cirrhosis and cirrhosis combined with HCC.

This study is designed as a hospital-based cross-sectional and randomized placebo-controlled intervention trial. One hundred and fifty patients with either cirrhosis or cirrhosis combined with HCC who meet the inclusion criteria will be recruited from Taichung General Veterans Hospital. One hundred patients will be randomly assigned to either the 1) placebo group (n = 25); 2) vitamin B-6 group; (50 mg/d, n = 25); 3) GSH group (500 mg/d, n = 25); or 4) vitamin B-6 (50 mg/d) plus GSH (500 mg/d) group (n = 25) for 3 mo. Data on demography, anthropometry and medical history will be collected. Patients with cirrhosis or cirrhosis combined with HCC will have fasting blood drawn in the clinics. Additionally, patients who participated in the intervention study will have blood drawn at month 0, 1, 2 and 3 during intervention period. Hematological, plasma vitamin B-6 status, GSH, inflammatory markers, homocysteine, cysteine, SAM, SAH, oxidative stress indicator, GSSG and GSH related antioxidant enzyme activities will be measured.

Hopefully, the results of this study could provide more pictures on the beneficial effects of vitamin B-6 and GSH supplementation on inflammatory responses, homocysteine, cysteine, the ratio of SAM/SAH, oxidative stress, GSSG and GSH related antioxidant enzyme activities in patients with cirrhosis and HCC.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 to 80 years old
2. patients are diagnosed as cirrhosis or cirrhosis combined with hepatocellular carcimoma

Exclusion Criteria:

1. patients are currently taking any nutrient supplements
2. patients with cardiac, renal, gastrointestinal or diabetic diseases
3. patients are currently taking any medication which will interfere with vitamin B-6 or glutathione metabolism〔i.e., phenobarbital, phenytoin, cycloserine, pyrazinamide, isoniazid, (thio)semicarbazide, hydramitrazine, phenelzine, carbidopa, levodopa, hydralazine, steroids and penicillamine)
4. patients are in pregnant or lactation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress marker (MDA concentation) | 3 months

SECONDARY OUTCOMES:
Glutathione related enzyme activities | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Bin Cheng, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan